CLINICAL TRIAL: NCT01170910
Title: Interest of Pulsatile Perfusion Preservation on Outcomes in Kidney Transplantation From Expanded Criteria Donors
Brief Title: Pulsatile Perfusion Preservation in Kidney Transplantation From Expanded Criteria Donors
Acronym: IMPULSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2009.550/3
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Chronic Renal Failure
Keywords: Chronic renal failure; Transplantation; Marginal kidney graft; Pulsatile perfusion machine
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Pulsatile Flow

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Static incubation (Other): If conservation in static incubation (group 1) is chosen by random selection, the transplant should be carried out while keeping the cold ischemic time (CIT) as short as possible (preferably less than 18 hours). Keep in mind that for reasons of homogeneity for result analysis and for conservation quality, it is recommended that kidneys in group 1 be conserved in University of Wisconsin (eg, UW, Belzer® or Viaspan®), IGL-1, or SCOT solution.
  Interventions: Procedure: Static incubation
- Pulsatile perfusion (Experimental): If conservation in a pulsatile perfusion machine (group 2) is chosen by random selection, the kidney will be placed in the perfusion machine within two hours and should be kept there at least 6 hours and 8 hours if possible, before being transplanted
  Interventions: Procedure: Pulsatile perfusion

INTERVENTIONS:
Procedure: Static incubation — Kidneys in this group are conserved in University of Wisconsin (eg, UW, Belzer® or Viaspan®), IGL-1, or SCOT solution before being transplanted.
  .
  Arms: Static incubation
Procedure: Pulsatile perfusion — Kidneys in this group are placed in the pulsatile perfusion machine(RM 3) within two hours and should be kept there at least 6 hours and 8 hours if possible, before being transplanted
  Arms: Pulsatile perfusion

SUMMARY:
Our hypothesis is that the Waters Medical® pulsatile perfusion machine (RM 3) is a way to improve delayed graft function (DGF) in marginal grafts, and some perfusion profiles (flow, pressure, resistance index, venous effluent pH) are correlated with better recovery of renal function (without dialysis during the first week after transplant).

Observation or Investigation Method Used :

The study is multicenter, prospective, open, controlled and randomized:grafts are divided into two parallel groups:

* group 1 corresponds to a conservation of grafts in static incubation
* group 2 corresponds to conservation using a pulsatile perfusion machine

Duration and Organizational Arrangements for Research :

The total duration of the study is planned for 36 months. This duration includes:

* an inclusion period that will last 24 months,
* the follow-up of recipient patients from the day of transplantation until twelve months after the operation

ELIGIBILITY:
Inclusion Criteria for marginal graft:

* donors over 60 years of age
* donors between 50 and 60 years of age with at least one of the following characteristics :

  * history of diabetes mellitus
  * history of high blood pressure
  * serum creatinine >1,5 mg/dL
  * death by stroke (haemorrhagic or thrombotic)

Inclusion criteria for recipient :

* patients registered on the kidney transplant waiting list likely to receive a marginal kidney
* immunized patients whose anti-HLA antibody specificities have been determined

Exclusion Criteria for recipient:

* pregnant or breastfeeding women
* people who have been incarcerated
* minors
* adults under guardianship
* people who are not affiliated with the French healthcare system
* people with HLA immunization whose HLA antibody specificities have not been determined

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Delayed graft function (DGF) rate defined as the need to resort to dialysis during the first week after transplantation. The main dialysis factors retained are hydrosodic and/or hyperkalemic overload. | First week after transplantation

SECONDARY OUTCOMES:
Evaluate improvement in the glomerular filtering rate | 12 months after transplantation
Evaluate the recourse to dialysis | 3 months following transplantation
Evaluate the proportion of functional grafts (which allows for renal purification without recourse to dialysis) | 12 months after transplantation
Evaluate patient survival | 12 months after transplantation
Stratify the analysis of regaining function and graft survival using Nyberg's classification in order to determine which risk groups would most benefit from pulsatile perfusion. | 12 months after transplantation
Identify perfusion profiles of the machine, which predict regaining renal function (absence of dialysis during the week after transplantation) and graft survival | 12 months after transplantation
Evaluate the medico-economic impact of each conservation strategy in the management of patients who will benefit from marginal grafts | 12 months after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Urologie et Chirurgie de la Tranplantation - Hôpital Edourad Herriot, Lyon, France

REFERENCES:
- [Derived] Tingle SJ, Thompson ER, Figueiredo RS, Moir JA, Goodfellow M, Talbot D, Wilson CH. Normothermic and hypothermic machine perfusion preservation versus static cold storage for deceased donor kidney transplantation. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD011671. doi: 10.1002/14651858.CD011671.pub3. PMID 38979743